CLINICAL TRIAL: NCT03292432
Title: Triggered Escalating Real-time Adherence Intervention to Promote Rapid HIV Viral Suppression Among Youth Living With HIV Failing Antiretroviral Therapy: The TERA Study
Brief Title: Triggered Escalating Real-time Adherence (TERA) Intervention
Acronym: TERA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 152; 5U24HD089880-02 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2021-01-08 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-10

CONDITIONS: HIV Infections
Keywords: Adherence, Medication
MeSH Terms: conditions — HIV Infections; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a Phase II, two-arm, randomized, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Standard of Care for adherence support at Site
  Interventions: Behavioral: Standard of Care (SOC)
- TERA Intervention (TERA) (Experimental): Triggered, escalating, real-time adherence (TERA) intervention for 12 weeks.
  Interventions: Behavioral: TERA Intervention (TERA)

INTERVENTIONS:
Behavioral: TERA Intervention (TERA) — A sequence of adherence support strategies implemented at care visits and as needed on the basis of EDM data. Components include: (1) remote education/preparation with an adherence coach conducted with VSee software (video conferencing) at site at baseline, week 4 and week 12; (2) one-way text alert at dose time when bottle has not yet been opened for that dosing window (users can disable this on request); (3) missed dose two-way outreach text asking "What's the plan?" which gets sent to both the participant's phone and a study phone; and (4) implementation of the coach-outreach (phone, text, remote counseling) triggered by missed doses or as a check-in to inquire about the well-being of the youth (once per week when no other contact with coach occurred the week prior).
  Arms: TERA Intervention (TERA)
Behavioral: Standard of Care (SOC) — Cell-phone reminders, patient-education, adherence planning (medication management), and checking-in on adherence at clinical care visits, as well as Viral load (VL) monitoring with patient feedback on VL, are used at sites. Less common, but available as a general service at some sites, on several websites, and at many pharmacies, youth may also receive text messages at dose times, for appointment reminders, and for refill reminders.
  Arms: Standard of Care (SOC)

SUMMARY:
Youth Living with HIV (YLWH) often face unique challenges achieving high and sustained rates of adherence to their antiretroviral therapy (ART). Poor adherence can lead to unsuppressed virus, more advanced HIV disease and poorer health outcomes, eventually exhausting treatment options. To date however, there are few demonstrated interventions for youth failing first line therapy. This study evaluated a novel intervention that used remote coaching through video enabled counseling sessions, an Electronic Dose Monitoring (EDM) pill bottle that notified an adherence coach when youth failed to open/close the device around dose time, and problem solving outreach by the coach in response to not dosing from the EDM. This intensive 'boot camp' strategy was implemented for 12 weeks followed by observation through 48 weeks.

DETAILED DESCRIPTION:
This was a Phase II, two-arm, randomized, open-label study. Eligible participants had failed ART therapy, defined as having a detectable plasma Human Immunodeficiency Virus - Type 1 Ribonucleic Acid (HIV-1 RNA) ≥200 copies/ml within 45 days of enrollment despite having been prescribed ART for at least 24 weeks. They could continue the same ART regimen or start a new once daily regimen. Participants were stratified by age (<18 vs. ≥18 years of age) and randomized in equal proportions to receive the study intervention (TERA) or standard of care (SOC), with no enrollment limits in each stratum. Target accrual was 120 participants to be enrolled over one year.

TERA was a time-limited (12 weeks) intervention approach that (a) used wireless electronic dose monitoring (EDM) to identify dose-times passing with no bottle opening, (b) sent a text asking about the delay, (c) evaluated response to the text and (d) initiated follow-up by an adherence coach depending on the response and if the bottle remained unopened for a designated period post dosing. Phone based outreach used problem solving discussion with an adherence coach, who could use an agreed-upon contact tree to reach the youth through other individuals. This "boot camp" strategy was used to unsettle or disrupt established non-adherence behaviors and factors promoting ongoing non-adherence.

Participants were followed for 48 weeks, with clinic visits at entry and weeks 4, 12, 24, 36 and 48. Audio computer assisted self-interviews (ACASI) were conducted every 12 weeks to collect information on adherence, motivation and skills, social support, mental and physical health functioning. Viral loads, medication and medical histories were also collected at each study visit.

The primary objective of the study was to compare HIV-virologic suppression (VLS) rates at 12 weeks. Secondary objectives included comparing VLS rates and EDM rates of ART adherence at 24, 36, and 48 weeks as well as patterns of adherence over time.

Major changes after the start of enrollment:

1. To address lower than anticipated enrollment, the requirement that participants be failing first line ART was dropped in Protocol Version 2.0 (May 9, 2018).
2. Accrual was closed before reaching the target enrollment of 120 participants on the recommendation of the Study Monitoring Committee (September 30, 2019).
3. Coronavirus disease of 2019 (COVID-19) Updates: On March 20, 2020, the TERA study suspended all study activities due to COVID-19. On May 5, 2020, sites were allowed to resume TERA study activities whenever their institution allowed human subjects research to resume. Participants were encouraged to return for their final Week 48 clinic visits.

At the time of the study pause, data collection for the Primary Outcome Measures was complete, so the analyses proposed in the original Statistical Analysis Plan were not affected. Follow-up for the Secondary Outcome Measures involving HIV-1 RNA measurements and adherence was incomplete, with 33% of participants still on study. Because of the possibility that participant behavior and adherence to ART would differ pre- and post-pandemic, and it would not be possible to collect HIV-1 RNA measurements within the required visit windows (sites were actively trying to keep patients from coming into care unless urgently needed), the Study Team decided to base analyses on data collected prior to the COVID-19 study pause. In addition, because the secondary virologic outcome measures were a combination of HIV-1 RNA levels and data completeness (classifying participants with no HIV-1 RNA measurement within the allowed visit window as "virologic failures"), the analysis population for these outcome measures only included participants with sufficient time on study to reach each study visit.

These changes were implemented on June 2, 2020 in a Letter of Amendment (LOA) to TERA Protocol Version 3.1. The LOA detailed three modifications due to COVID-19 study visit suspension, but did not affect the existing protocol:

1. Extension of Week 48 visit window through the end of data collection (October 12, 2020) for participants on-study as of March 20, 2020, due to COVID-19 study suspension.
2. Changed all secondary outcome measures to apply only to data collected prior to COVID-19 study suspension on March 20, 2020. Only participants who had been on study long enough to reach the Week 24, 36 or 48 study visits were included in the analyses.
3. Virtual/remote site monitoring was implemented for all remaining site monitoring visits.

On September 24, 2020, the Study Team released a memo to the sites extending the date for the Week 48 study visit to October 12, 2020.

Results for secondary outcome measures 3 to 8 are based on the pre COVID-19 study pause database as of March 20, 2020.

Results for secondary outcome measures 9 and 10 are based on the complete study database as of October 12, 2020.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of HIV-1 Infection as documented in the participant's medical record by at least two of the following criteria:

   * Reactive HIV screening test result with an HIV antibody or HIV antibody/antigen-based, Food and Drug Administration (FDA)-licensed assay followed by a positive supplemental assay (e.g., HIV-1 Western Blot, HIV-1 indirect immunofluorescence, HIV-1/HIV-2 discriminatory immunoassay);
   * Plasma HIV-1 quantitative ribonucleic acid (RNA) assay >1,000 copies/mL;
   * Positive HIV-1 deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assay; or
   * Positive plasma HIV-1 RNA qualitative assay
2. Participant aware of his or her HIV infection, as determined by site staff
3. Documented plasma HIV-1 RNA plasma ≥200 copies/mL within 45 days of the date of the enrollment visit
4. Prescribed antiretroviral therapy for at least 24 weeks or more prior to documented plasma HIV-1 RNA plasma ≥200 copies/mL.
5. Prescribed a once-daily (one or more pills once a day) ART regimen with at least two active agents (per clinician judgment or genotype evidence) at enrollment
6. Able to communicate in spoken and written English
7. Currently has a cellular phone that is also able to send and receive text messages
8. Willing and able to provide at least one additional contact phone number (preferably two) to contact participant
9. Able and willing to provide written informed assent/consent and able to obtain written parental or guardian permission (if required as specified by the site, by state law, and/or Institutional Review Board policy, and detailed in each site's Protocol Implementation Plans) to be screened for and to enroll in this study

Exclusion Criteria:

1. Gross cognitive limitations, acute emotional instability, or medical or mental health illness that in the opinion of site personnel would impair the individual's ability to provide informed consent and/or interfere with the protocol's objectives
2. Concurrent participation in interventional studies addressing adherence unless approved in advance by study team
3. Positive pregnancy test at the time of enrollment. If participant becomes pregnant while on study, they may continue on study
4. Currently using or planning to use an electronic dose monitoring and reminder device outside of the study

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 89 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: K. Rivet Amico, PhD, Principal Investigator — University of Michigan School of Public Health; Michael Hudgens, PhD, Study Director — University of North Carolina, Chapel Hill; Aditya H Gaur, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (8):
  - University of Colorado Denver Children's Hospital Colorado, Aurora, Colorado
  - Broward Health Childrens Diagnostic and Treatment Center (CDTC), Fort Lauderdale, Florida
  - University of Florida Center for HIV/AIDS, Research, Education & Service, Jacksonville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Wayne State University School of Medicine, Detroit, Michigan
  - Bronx-Lebanon Hospital Center, The Bronx, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amico KR, Dunlap A, Dallas R, Lindsey J, Heckman B, Flynn P, Lee S, Horvath K, West Goolsby R, Hudgens M, Filipowicz T, Polier M, Hill E, Mueller Johnson M, Miller J, Neilan A, Ciaranello A, Gaur A. Triggered Escalating Real-Time Adherence Intervention to Promote Rapid HIV Viral Suppression Among Youth Living With HIV Failing Antiretroviral Therapy: Protocol for a Triggered Escalating Real-Time Adherence Intervention. JMIR Res Protoc. 2019 Mar 18;8(3):e11416. doi: 10.2196/11416. PMID 30882360
- [Derived] Lindsey JC, Hudgens M, Gaur AH, Horvath KJ, Dallas R, Heckman B, Mueller Johnson M, Amico KR. Electronic Dose Monitoring Device Patterns in Youth Living With HIV Enrolled in an Adherence Intervention Clinical Trial. J Acquir Immune Defic Syndr. 2023 Mar 1;92(3):231-241. doi: 10.1097/QAI.0000000000003126. PMID 36730762
- [Derived] Amico KR, Crawford J, Ubong I, Lindsey JC, Gaur AH, Horvath K, Goolsby R, Mueller Johnson M, Dallas R, Heckman B, Filipowicz T, Polier M, Rupp BM, Hudgens M. Correlates of High HIV Viral Load and Antiretroviral Therapy Adherence Among Viremic Youth in the United States Enrolled in an Adherence Improvement Intervention. AIDS Patient Care STDS. 2021 May;35(5):145-157. doi: 10.1089/apc.2021.0005. PMID 33960843

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 sites in the United States between April 12, 2018 and September 30, 2019.
Pre-assignment Details: Participants were stratified by age (< 18 years vs. >= 18 years) and randomized equally to the TERA intervention and Standard of Care. One participant was randomized but never started a behavioral intervention as site closed before any data collected.
Period: Overall Study
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Started (Number enrolled) | 46 | 43
Started Study Intervention (Number starting intervention) | 45 | 43
Completed | 31 | 32
Not Completed | 15 | 11
Not completed — Lost to Follow-up | 11 | 8
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Site closed before any data collected | 1 | 0

BASELINE CHARACTERISTICS:
Population: Includes participants who started study intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA) | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Median (Full Range); unit: years] | 22.1 [16.5 to 24.8] | 22.3 [13.7 to 24.8] | 22.2 [13.7 to 24.8]
Age, Customized [Count of Participants; unit: Participants]
  13 - 17 years | 5 | 4 | 9
  18 - 21 years | 16 | 13 | 29
  22 - 25 years | 24 | 26 | 50
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 19 | 21 | 40
    Male | 26 | 22 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 41 | 34 | 75
  Unknown or Not Reported | 0 | 4 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 34 | 74
  White | 2 | 0 | 2
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 43 | 88
Mode of transmission [Count of Participants; unit: Participants]
  Horizontal transmission | 24 | 25 | 49
  Vertical transmission | 21 | 18 | 39
Plasma Human Immunodeficiency Virus - Type 1 Ribonucleic Acid (HIV-1 RNA) [Count of Participants; unit: Participants]
  200 - <400 copies/mL | 4 | 6 | 10
  400 - <10,000 copies/mL | 25 | 21 | 46
  10,000 - <50,000 copies/mL | 9 | 5 | 14
  >= 50,000 copies/mL | 7 | 11 | 18
Cluster of differentiation 4 (CD4) cell count [Count of Participants; unit: Participants]
  < 200 cells/mm^3 | 4 | 11 | 15
  200 - < 500 cells/mm^3 | 16 | 13 | 29
  500 - < 1000 cells/mm^3 | 22 | 17 | 39
  >= 1000 cells/mm^3 | 2 | 2 | 4
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus - Type I Ribonucleic Acid (HIV-1 RNA) Levels Less Than (<) 50 Copies/mL at Week 12
Description: Participants with HIV-1 RNA < 50 copies/mL within the week 12 window (+/- 14 days) are classified as successes. Participants with HIV-1 RNA >= 50 copies/mL or with no HIV-1 RNA measurement within the week 12 window are classified as failures.
Time Frame: 12 weeks post enrollment
Population: Includes participants who started study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 43
Percentage of participants | 24.4 | 20.9
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Test type: Superiority; p = 0.80, Fisher Exact; Risk Difference (RD) = -3.5, 95% CI 2-sided [-21.8 to 15.2] — Risk difference reflects percentage of participants achieving HIV-1 RNA < 50 copies/mL in TERA arm minus SOC arm

2. Primary Outcome: Percentage of Participants With HIV-1 RNA < 200 Copies/mL at Week 12
Description: Participants with HIV-1 RNA < 200 copies/mL within the week 12 window (+/- 14 days) are classified as successes. Participants with HIV-1 RNA >= 200 copies/mL or with no HIV-1 RNA measurement within the week 12 window are classified as failures.
Time Frame: 12 weeks post enrollment
Population: Includes participants who started study intervention
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 43
Percentage of participants | 35.6 | 34.9
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Test type: Superiority; p > 0.99, Fisher Exact; Risk Difference (RD) = -0.7, 95% CI 2-sided [-20.9 to 19.6] — Risk difference reflects percentage of participants achieving HIV-1 RNA < 200 copies/ml in TERA arm minus SOC arm

3. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Weeks 24, 36 and 48
Description: Participants with HIV-1 RNA < 50 copies/mL within each week window (+/- 28 days) are classified as successes. Participants with HIV-1 RNA >= 50 copies/mL or who had the opportunity to reach the study visit week and with no HIV-1 RNA measurement within the week window are classified as failures.
Time Frame: 24, 36 and 48 weeks post enrollment
Population: Includes participants who started study intervention and with the opportunity to reach the targeted study visit prior to the Coronavirus Disease 2019 (COVID-19) study pause on March 20, 2020
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 43
Percentage of participants
  Week 24: number analyzed (Participants) | 44 | 43
  Week 24 | 36.4 | 23.3
  Week 36: number analyzed (Participants) | 32 | 36
  Week 36 | 15.6 | 19.4
  Week 48: number analyzed (Participants) | 25 | 29
  Week 48 | 24.0 | 27.6
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages at Week 24; Test type: Superiority; p = 0.24, Fisher Exact; Risk Difference (RD) = -13.1, 95% CI 2-sided [-32.1 to 7.2] — Risk difference reflects percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 in TERA arm minus SOC arm
Statistical Analysis 2: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages at Week 36; Test type: Superiority; p = 0.76, Fisher Exact; Risk Difference (RD) = 3.8, 95% CI 2-sided [-16.0 to 22.6] — Risk difference reflects percentage of participants with HIV-1 RNA < 50 copies/mL at Week 36 in TERA arm minus SOC arm
Statistical Analysis 3: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages at Week 48; Test type: Superiority; p > 0.99, Fisher Exact; Risk Difference (RD) = 3.6, 95% CI 2-sided [-21.8 to 27.4] — Risk difference reflects percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 in TERA arm minus SOC arm

4. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 200 Copies/mL at Weeks 24, 36 and 48
Description: Participants with HIV-1 RNA < 200 copies/mL within each week window (+/- 28 days) are classified as successes. Participants with HIV-1 RNA >= 200 copies/mL or who had the opportunity to reach the study visit week and with no HIV-1 RNA measurement within the week window are classified as failures.
Time Frame: 24, 36 and 48 weeks post enrollment
Population: Includes participants who started study intervention and with the opportunity to reach the targeted study visit prior to the COVID-19 study pause on March 20, 2020
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 43
Percentage of participants
  Week 24: number analyzed (Participants) | 44 | 43
  Week 24 | 40.9 | 27.9
  Week 36: number analyzed (Participants) | 32 | 36
  Week 36 | 21.9 | 33.3
  Week 48: number analyzed (Participants) | 25 | 29
  Week 48 | 32.0 | 27.6
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages at Week 24; Test type: Superiority; p = 0.26, Fisher Exact; Risk Difference (RD) = -13.0, 95% CI 2-sided [-32.7 to 7.3] — Risk difference reflects percentage of participants with HIV-1 RNA < 200 copies/mL at Week 24 in TERA arm minus SOC arm
Statistical Analysis 2: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages at Week 36; Test type: Superiority; p = 0.42, Fisher Exact; Risk Difference (RD) = 11.5, 95% CI 2-sided [-11.2 to 32.8] — Risk difference reflects percentage of participants with HIV-1 RNA < 200 copies/mL at Week 36 in TERA arm minus SOC arm
Statistical Analysis 3: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages at Week 48; Test type: Superiority; p = 0.77, Fisher Exact; Risk Difference (RD) = -4.4, 95% CI 2-sided [-29.5 to 20.7] — Risk difference reflects percentage of participants with HIV-1 RNA < 200 copies/mL at Week 48 in TERA arm minus SOC arm

5. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 200 Copies/mL at 12 Weeks and Maintained Through 48 Weeks
Description: Participants are classified as successes if both the week 12 (+/- 14 days) and week 48 (+/- 28 days) HIV-1 RNA measurements are < 200 copies/mL and at least one of the week 24 (+/- 28 days) or week 36 (+/- 28 days) HIV-1 RNA measurements is < 200 copies/mL. Otherwise, the participant is classified as a failure.
Time Frame: 48 weeks post enrollment
Population: Includes participants who started study intervention and with the opportunity to reach the Week 48 visit prior to the COVID-19 study pause on March 20, 2020
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 25 | 29
Percentage of participants | 8.0 | 13.8
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Test type: Superiority; p = 0.67, Fisher Exact; Risk Difference (RD) = 5.8, 95% CI 2-sided [-14.6 to 25.3] — Risk difference reflects percentage of participants with HIV-1 RNA < 200 copies/mL at Week 12 and maintained to Week 48 in TERA arm minus SOC arm

6. Secondary Outcome: Percentage of Days With Dose Taken From Weeks 0-12, >12-24, >24-36 and >36-48
Description: For each participant and each 12-week period, the percentage is calculated as the number of days with dose taken divided by the number of days with data reported in the Electronic Monitoring Device (EDM).
Time Frame: Enrollment through 48 weeks
Population: Includes participants who started study intervention and with data reported in the adherence EDM up to the COVID-19 pause on March 20, 2020
Measure: Median (Inter-Quartile Range); unit: Percentage of days with dose taken
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 42
Percentage of days with dose taken
  Weeks 0 - 12 | 41.0 [20.5 to 59.0] | 72.1 [46.5 to 89.2]
  Weeks >12 - 24: number analyzed (Participants) | 45 | 39
  Weeks >12 - 24 | 14.3 [1.2 to 32.1] | 40.5 [10.7 to 70.2]
  Weeks >24 - 36: number analyzed (Participants) | 41 | 38
  Weeks >24 - 36 | 2.4 [0.0 to 14.3] | 17.2 [2.3 to 40.5]
  Weeks >36 - 48: number analyzed (Participants) | 27 | 31
  Weeks >36 - 48 | 1.2 [0.0 to 7.4] | 1.2 [0.0 to 30.0]
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages of doses taken from Weeks 0 -12; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentage of doses taken from Weeks >12 to 24; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentage of doses taken from Weeks >24 to 36; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentage of doses taken from Weeks >36 to 48; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Days With Dose Taken Within Defined Acceptable Window (+/- 4 Hours) From Weeks 0-12, >12-24, >24-36 and >36-48
Description: For each participant and each 12-week period, the percentage is calculated as the number of days with dose taken within acceptable window divided by the number of days with data reported in the EDM.
Time Frame: Enrollment through 48 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percentage of days dose taken on time
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 42
Percentage of days dose taken on time
  Weeks 0 - 12 | 21.4 [8.4 to 38.6] | 62.7 [30.1 to 84.3]
  Weeks >12 - 24: number analyzed (Participants) | 45 | 39
  Weeks >12 - 24 | 7.1 [0.0 to 16.7] | 27.4 [7.1 to 57.1]
  Weeks >24 - 36: number analyzed (Participants) | 41 | 38
  Weeks >24 - 36 | 2.4 [0.0 to 9.5] | 10.7 [0.0 to 35.7]
  Weeks >36 - 48: number analyzed (Participants) | 27 | 31
  Weeks >36 - 48 | 0.0 [0.0 to 4.8] | 1.2 [0.0 to 22.5]
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentage of doses taken on time from Weeks 0 - 12; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentage of doses taken on time from Weeks >12 - 24; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of percentages of doses taken on time from Weeks >24 - 36; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — p-value equal to a priori threshold for statistical significance
Statistical Analysis 4: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of doses taken on time from Weeks >36 - 48; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Incidence Rate of 7-day Gaps Between Dosing for Weeks 0-12, >12-24, >24-36 and >36-48
Description: For each participant, the incidence rate during each 12 week interval is calculated as the ratio of the number of 7-day gaps between doses relative to the number of weeks with data reported, times 12. Consecutive gaps of more than 7 days increase the gap count by one, e.g., missing 20 days counts as 2 gaps.
Time Frame: Enrollment through 48 weeks
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 45 | 42
Ratio
  Weeks 0 - 12 | 4.17 [3.61 to 4.82] | 1.66 [1.31 to 2.11]
  Weeks >12 - 24: number analyzed (Participants) | 45 | 39
  Weeks >12 - 24 | 6.91 [6.16 to 7.75] | 4.43 [3.81 to 5.15]
  Weeks >24 - 36: number analyzed (Participants) | 41 | 38
  Weeks >24 - 36 | 8.19 [7.28 to 9.21] | 6.65 [5.84 to 7.57]
  Weeks >36 - 48: number analyzed (Participants) | 27 | 31
  Weeks >36 - 48 | 9.54 [8.37 to 10.89] | 8.81 [7.76 to 10.00]
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of incidence rates from Weeks 0 - 12; Test type: Superiority; p < 0.001, Chi-squared; Pearson Chi-square test from generalized linear model with Poisson link; Risk Ratio (RR) = 2.51, 95% CI 2-sided [1.90 to 3.33] — Risk ratio for SOC arm relative to TERA arm
Statistical Analysis 2: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of incidence rates from Weeks >12 - 24; Test type: Superiority; p < 0.001, Chi-squared; Pearson Chi-square test from generalized linear model with Poisson link; Risk Ratio (RR) = 1.56, 95% CI 2-sided [1.29 to 1.89] — Risk ratio for SOC arm relative to TERA arm
Statistical Analysis 3: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of incidence rates from Weeks >24 - 36; Test type: Superiority; p = 0.020, Chi-squared; Pearson Chi-square test from generalized linear model with Poisson link; Risk Ratio (RR) = 1.23, 95% CI 2-sided [1.03 to 1.47] — P-value from Pearson Chi-square test from generalized linear model with Poisson link
Statistical Analysis 4: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Comparison of incidence rates from Weeks >36 - 48; Test type: Superiority; p = 0.39, Chi-squared; Pearson Chi-square test from generalized linear model with Poisson link; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.90 to 1.30] — Risk ratio for SOC arm relative to TERA arm

9. Other Pre Specified Outcome: Percentage of Participants With HIV-1 RNA < 200 Copies/mL at Week 48
Description: Participants with HIV-1 RNA < 200 copies/mL at Week 48 are classified as successes. Participants with HIV-1 RNA >= 200 copies/mL or with no HIV-1 RNA measurement after 44 weeks follow-up are classified as failures.
Time Frame: 48 weeks post enrollment
Population: Includes participants who started study intervention. Excludes participants who died from non-HIV-related causes before Week 48.
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 43 | 43
Percentage of participants | 23.3 | 25.6
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Test type: Superiority; p > 0.99, Fisher Exact; Risk Difference (RD) = 2.3, 95% CI 2-sided [-16.4 to 21.1] — Risk difference reflects percentage of participants achieving HIV-1 RNA < 200 copies/mL in TERA arm minus SOC arm

10. Other Pre Specified Outcome: Percentage of Participants With HIV-1 RNA < 200 Copies/mL at 12 Weeks and Maintained Through 48 Weeks
Description: as for outcome 5
Time Frame: 12, 24, 36, and 48 weeks post enrollment
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
Number analyzed (Participants) | 43 | 43
Percentage of participants | 7.0 | 11.6
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs TERA Intervention (TERA); Test type: Superiority; p = 0.71, Fisher Exact; Risk Difference (RD) = 4.7, 95% CI 2-sided [-9.0 to 19.4] — Risk difference reflects percentage of participants achieving sustained virologic control in TERA arm minus SOC arm

ADVERSE EVENTS:
Time Frame: From study entry to study completion (approximately 48 weeks)
Description: In addition to collection of serious adverse events, the study collected 'Untoward events' of Grade 3 or higher and related to the study. Untoward events were defined as unexpected occurrences involving study participants, study staff, or the community where the study was taking place, that may reasonably be judged as related to study procedures and that led to harm, distress, or increased risk of harm or distress, but that did not otherwise meet the definition of an adverse event.
Arm/Group | Standard of Care (SOC) | TERA Intervention (TERA)
All-Cause Mortality (participants affected / at risk) | 2/45 | 1/43
Serious Adverse Events (participants affected / at risk) | 3/45 | 4/43
Other Adverse Events (participants affected / at risk) | 0/45 | 2/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=45) | TERA Intervention (TERA) (N=43)
Cardiac event (Cardiac disorders) | 1 (1) | 0 (0) — Resulted in death
Esophageal candidiasis and pelvic inflammatory disease (Infections and infestations) | 1 (1) | 0 (0) — Resulted in hospitalization
Gunshot wound to head (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Resulted in death
Axillary abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax acute recurrent with shortness of breath, hypoxia and hypokalemia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HSV proctitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Facial cellulitis and MRSA positive wound of the tragus (Infections and infestations) | 0 (0) | 1 (1)
AIDS (Infections and infestations) | 0 (0) | 1 (1) — Resulted in death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=45) | TERA Intervention (TERA) (N=43)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Accrual was closed before reaching the targeted enrollment of 120 participants. Study visits were paused on March 20, 2020 due to the outbreak of COVID-19, interrupting systematic collection of secondary outcome measures. Statistical comparisons between arms therefore had lower than anticipated power to detect differences. For EDM data, the time the device was opened can only be assumed to correspond with when the participant took their antiretroviral dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT03292432/SAP_000.pdf
  • Study Protocol: Protocol Version 3.1 (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT03292432/Prot_001.pdf
  • Study Protocol: Letter of Amendment to Study Protocol Version 3.1 (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT03292432/Prot_002.pdf